CLINICAL TRIAL: NCT05151666
Title: Assessing the Impact of Intra-dialytic Exercise Regimen on Depression Scores
Brief Title: Exercise in Dialysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Initially the study failed to start due to Covid concerns. As this is an immunocompromised patient population, this concern has persisted and study initiation was further complicated by a demographic and availability change in research team members.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-00989
Record Dates: First submitted 2021-12-01; First posted 2021-12-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Depression
Keywords: Hemodialysis
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Single arm pre-post intervention study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodialysis Patients (Experimental)
  Interventions: Other: Sunny Health & Fitness Magnetic Mini Exercise Pedal Cycle - SF-B020026 Gray

INTERVENTIONS:
Other: Sunny Health & Fitness Magnetic Mini Exercise Pedal Cycle - SF-B020026 Gray — The intervention will be that the patient cycles in a sitting position within the first 2 hours of hemodialysis treatment for 15-60 minutes/as tolerated, either intermittent/continuous duration. - Graded duration will increase every 2 weeks. This will be supervised by a dialysis nurse as per the schedule of study assessments.

SUMMARY:
The purpose of the proposed clinical trial is to support intradialytic pedal cycling exercise as an intervention and show its effect on depression and how there is a need for more programs to support this. This is an exploratory single arm study. These patients will be cycling during dialysis treatment by using a graded duration model. Even though patients on hemodialysis (HD) have an increased life span due to renal replacement therapy, exercise can have a remarkable effect on their ability to perform daily activities. Dialysis has been shown to reduce self-confidence, increase social isolation, and cause feelings of disappointment in the future. This population faces mental and psychological stress due to the disease burden. Short-term supervised cycling programs while patients are receiving dialysis have been reported to induce systematic improvements for depression and anxiety. Exercise during hemodialysis is an effective way to reduce depressive symptoms without using pharmacologic measures.

Data for each patient will be collected at each dialysis treatment using a unique patient identifier. The data that will be collected include duration of exercise (intermittent or continuous), any complications during HD, vital signs while cycling every 30 minutes, and how they state they feel after cycling. The measurable outcome will be depression scores. The tool that will be used for this project is the Beck Depression Inventory (BDI). The patient will complete the BDI assessment on week 1 (pre intervention as baseline) and then on week 10 (post intervention).

ELIGIBILITY:
Inclusion Criteria:

1. greater than 18 years of age
2. male or female
3. ESKD on maintenance hemodialysis for 3 consecutive months
4. adequate dialysis clearances (Kt/V greater than 1.2),
5. able to participate in exercise program based on nephrologist evaluation
6. able to provide written informed consent for participation,
7. Compliance with dialysis treatment regimen (attended 75% of ordered dialysis treatments in the last 3 months.

Exclusion Criteria:

1. less than 18 years old
2. on hemodialysis for < 3 consecutive months
3. acute Kidney Injury diagnosis
4. patients deemed clinically unstable by Nephrologist
5. active foot ulcer
6. unable to provide written consent
7. refusal of participation
8. lower limb amputations
9. patients with dementia or severe cognitive impairment
10. patients with Psychiatric disorders (who are not treated and unstable)
11. pregnancy
12. myocardial infarction in the last 6 months
13. uncontrolled diabetes
14. patients on chronic Midodrine therapy for intradialytic blood pressure support.
15. deep vein thrombosis
16. symptomatic peripheral vascular disease and/or recent lower extremities vascular intervention (i.e. bypass)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-02 (Estimated); Primary Completion 2024-03-11 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory (BDI) Score | Week 1, Week 10
  BDI is a 21-item self-report scale designed to measure the severity of depressive symptoms. Each item is scored 0-3. The total score range is 0-63; the higher the score, the more severe the depression. A score > 40 indicates extreme depression.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Masani, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Dialysis Center of Bethpage, Bethpage, New York
  - NYU Winthrop Dialysis Center - Outpatient, Mineola, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Naveed.Masani@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.